CLINICAL TRIAL: NCT04795128
Title: A Phase I Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 in Subjects With Hematologic Malignancy
Brief Title: A Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 in Subjects With Hematologic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI322A103
Record Dates: First submitted 2021-02-26; First posted 2021-03-12 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI322 (Other): Single arm
  Interventions: Biological: IBI322

INTERVENTIONS:
Biological: IBI322 — Recombinant anti-human CD47/PD-L1 bispecific antibody injection

SUMMARY:
This is a phase I study evaluating the safety, tolerability and preliminary efficacy of IBI322 in subjects with hematologic malignancies who have failed standard treatment.

DETAILED DESCRIPTION:
This Phase 1a/1b study will be conducted to evaluate the safety, tolerability, PK, PD, immunogenicity, and preliminary antitumor activity of IBI322 in China. Phase 1a is a dose escalation and plans to enroll approximately 39-102 subjects with hematologic malignancies who have failed standard treatments. Phase 1b is a dose expansion and plans to enroll approximately 80 subjects with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed hematologic malignancy who failed the standard treatment
2. At least one evaluable lesion
3. Male or female 18 to 75 years old
4. Eastern Cooperative Oncology Group Performance Status Performance Status (ECOG PS) 0-2
5. Must have adequate organ function

Exclusion Criteria:

1. Previous exposure to any anti-CD47 monoclonal antibody, SIRPα antibody, or CD47/SIRPα recombinant protein
2. Previous exposure to chimeric antigen receptor T cell immunotherapy (CAR-T)
3. Subjects participating in another interventional clinical study, except for: observational (non-interventional) clinical studies or survival follow-up phase of interventional studies
4. Use of anticoagulants and/or aspirin, or other non-steroidal anti-inflammatory drugs within 2 weeks prior to study start
5. A history of blood transfusion within 2 weeks prior to study start

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Number of treatment related AEs | Up to 90 days post last dose
  Safety
Number of patients with response | Last patient enrolled +24 weeks
  Preliminary Efficacy

SECONDARY OUTCOMES:
PK Parameters: The area under the curve (AUC) | Up to 90 days post last dose
  Safety and Preliminary Efficacy
PK Parameters: Maximum concentration (Cmax) | Up to 90 days post last dose
  Safety and Preliminary Efficacy
PK Parameters: Half-life (t1/2) | Up to 90 days post last dose
  Safety and Preliminary Efficacy
PK Parameters: Clearance (CL) | Up to 90 days post last dose
  Safety and Preliminary Efficacy
PK Parameters: Volume of Distribution (V) | Up to 90 days post last dose
  Safety and Preliminary Efficacy
Positive Rate of ADA and Nab | Up to 90 days post last dose
  Safety and Preliminary Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: WenBin Qian, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang, China